CLINICAL TRIAL: NCT03556306
Title: Unexpected Intraoperative Findings and Complications in Bariatric Surgery
Brief Title: Intraoperative Findings and Complications in Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Hospital General Tlahuac (Other Government)
Responsible Party: Principal Investigator, CARLOS ZERRWECK LOPEZ, Professor, Hospital General Tlahuac
Other Study IDs: 09-CEI-001-20160404; 212-010-22-17 (Registry Identifier: Institutional Register)
Record Dates: First submitted 2018-05-31; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Bariatric Surgery; Complication of Surgical Procedure; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — The gastric bypass ("simplified technique") was performed in an antecolic fashion, with a calibrated 2 cm gastro-jejunal anastomosis (linear stapler); biliary and alimentary limbs measured 70 and 150 cm respectively [17] . Mesenteric defects were closed and the omentum divided. The sleeve gastrectomy was performed at 5-6 cm from the pylorus over a 36 Fr. bougie, with oversuture of the staple line (2-0 polypropylene). Methylene blue test and the use of drains were done routinely.
  Other Names: Laparoscopic gastric bypass; Sleeve gastrectomy; Revisional surgery

SUMMARY:
Retrospective study with patients submitted to bariatric surgery between 2013 and 2016 at a single Institution. The objective was to analyze the incidence and causes of unexpected intraoperative findings and complications, change in surgical plan, extra surgeries and procedure interruption. All operative information was collected prospectively and aimed to describe any of the previous situations. Secondarily, a morbidity analysis was performed, correlating intraoperative complications with postoperative complications and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patient submitted to bariatric surgery
* All patients met the guidelines defined by the National Institutes of Health (NIH) consensus: BMI equal or greater to 40kg/m2 or BMI 35 - 40 kg/m2 with some comorbidity

Exclusion Criteria:

* Patients with incomplete surgery data sheet and those subject to another type of bariatric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with obesity submitted to bariatric surgery (LGBP, LSG, and revisional surgery) in a single institution between January 2013 and March 2016.
Sampling Method: Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative Complications | During surgical time
  yes/no
Intraoperative unexpected findings, change in surgical technique, surgery interruption | During surgical time
  yes/no

SECONDARY OUTCOMES:
Postoperative complications | 0-30 days
  (yes/no) (minor/major)
Length of Hospital Stay | 0-30 days
  Days

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS ZERRWECK, MD, Study Director — The Obesity Clinic at Hospital General Tlahuac; Paul Joo, MD, Principal Investigator — The Obesity Cklinic at Hospital General Tlahuac
Locations (1):
- The Obesity Clinic at Hospital General Tlahuac, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided